CLINICAL TRIAL: NCT06570330
Title: Assessing the Impact of Daily Supplementation of a Multi - Human Milk Oligosaccharide (HMO) Formulation on Adult Gut Microbiome Health
Brief Title: Adult HMO Supplementation and the Gut Microbiome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seeding, Inc DBA Tiny Health (Industry)
Collaborators: Mellitas Health Foods, LLC (DBA Layer Origin Nutrition) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: LO_12186.01
Record Dates: First submitted 2024-08-20; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - SuperHMO (Experimental): The investigation product is commercially available and is marketed as SuperHMO Prebiotic Mix with 5 HMOs. This product is a dietary supplement which contains five major types of human milk oligosaccharides includes 2'-Fucosyllactose (2'-FL), Lacto-N-tetraose (LNT), Lacto-N-neotetraose (LNnT), 6'-Sialyllactose (6'SL), and 3'-Sialyllactose (3'SL). SuperHMO is designed to boost the number and variety of beneficial bacteria in the gut by feeding them with five different kinds of human milk oligosaccharide prebiotics. This product does not contain any flavoring, colorants, preservatives or fillers. Each bottle contains 118 grams of the mix, 28 servings, with 4.2 grams per serving (2 scoops).
  Study participants will be instructed to take 1 scoop (2.1 g) per day for the first five days and increase to 2 scoops (4.2g) per day for days 6-30, the formulation can be dissolved in their beverage of choice and taken at any time of the day, with or without food.
  Interventions: Dietary Supplement: SuperHMO
- Control (Placebo Comparator): Control participants will receive a commercially available maltodextrin, NOW Sports Nutrition, Non-GMO corn Maltodextrin, Rapid Absorption. The composition and absorption properties are similar to the investigational product and will be given in the same dosage (2.1g/day for days 1-5 and increasing to 4.2 g/day for days 6-30) and route of administration as the investigational product. The use of maltodextrin as a comparator in prebiotic supplementation in human trials is well-documented.
  Interventions: Dietary Supplement: Non-GMO corn Maltodextrin, Rapid Absorption

INTERVENTIONS:
Dietary Supplement: SuperHMO — Super HMO Prebiotic Mix: five major types of human milk oligosaccharides including 2'-Fucosyllactose (2'-FL), Lacto-N-tetraose (LNT), Lacto-N-neotetraose (LNnT), 6'-Sialyllactose (6'SL), and 3'-Sialyllactose (3'SL)
  Arms: Intervention - SuperHMO
Dietary Supplement: Non-GMO corn Maltodextrin, Rapid Absorption — he composition and absorption properties are similar to the investigational product and will be given in the same dosage (2.1g/day for days 1-5 and increasing to 4.2 g/day for days 6-30) and route of administration as the investigational product.
  Arms: Control

SUMMARY:
The goal of this study is to assess the impact of Layer Origin's SuperHMO prebiotic formulation on the healthy adult gut microbiome. Over the course of 30 days, intervention participants will take SuperHMO prebiotic formulation daily. Control participants will take a placebo daily. We will measure all participants' gut microbiome using a gut health test before taking SuperHMO prebiotic or placebo and after 30 days of taking the supplement. We hypothesize that taking the SuperHMO prebiotic will improve gut health measurements such as the potential to produce short-chain fatty acids.

DETAILED DESCRIPTION:
The investigators will enroll 24 healthy, adult volunteers into this double-blinded, randomized, placebo-controlled trial. Upon confirmation of eligibility and documentation of informed consent, the participants will be randomized to either SuperHMO (Layer Origin, 53% 2'FL, 15% LNT, 14%LNnT, 12% 6'SL, 6% 3'SL) prebiotic formulation at a dosage of (4.2 g/day) or placebo (maltodextrin, 4.2 g/day), self-administered at home and taken as a liquid solution in a beverage of choice by mouth once daily for 30 days. Participants will take a baseline survey at the beginning of the study and an exit survey at the end of the study assessing their current health, health history, diet, current and past supplement and medication use, and any GI symptoms or bowel irregularities. Participants will additionally take a baseline microbiome sample before beginning the daily regimen of taking the supplement or placebo for 30 days. At the end of the study, participants will take another microbiome sample and an exit survey to report changes to gut health, overall health, diet, and any adverse reactions. Gut microbiome outcomes will be analyzed both intra-individually, as a before and after comparison, and inter-individually to compare intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants are between the ages of 18 and 40.

Exclusion Criteria:

* Participants cannot have taken prebiotic or probiotic supplements within 6 months of starting study. This includes prebiotic or probiotic powder or supplements with prebiotic or probiotic addition or multivitamin with probiotic addition. This does not include food with live probiotics in it like yogurt or kefir.

  * Participants must not be pregnant or breastfeeding or trying to conceive within the study period.
  * Participants must be residents of the United States with US postal service.
  * Participants cannot have the following existing health conditions:

    * Pre-existing gut conditions (IBD, Celiac's disease, Crohn's disease, SIBO)
    * Immune or auto-immune conditions (Type 1 Diabetes, human immunodeficiency virus (HIV))
  * Participants cannot be lactose intolerant or have an allergy to dairy products.
  * Participants are excluded if they have received results from an at home microbiome stool test in the past 6 months. This does not include clinical workup such as culture or pathogen testing.
  * Participants must agree not to take another prebiotic or probiotic supplement or an at-home test over the study period.
  * Participants must have no known major dietary changes upcoming.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Quantitative changes in the relative abundance of key bacterial taxa | 30 days
  The investigators will specifically measure the difference in Bifidobacterium spp., Akkermansia spp., Eubacterium rectale-Clostridium Coccoides group, and Faecalibacterium prausnitzii, at baseline and at 30 days.
Detection of presence of specific HMO digestion genes | 30 days
  Comparing baseline and again after 30 days of taking the study product to assess potential changes in HMO metabolism by the gut microbiota.
Assess Changes in the diversity metrics of the Gut Microbiome | 30 days
  Measuring the change in alpha diversity (e.g., Shannon index) and beta diversity metrics (e.g., Bray-Curtis dissimilarity) to evaluate overall microbial diversity and community structure shifts between baseline and at 30 days.
Evaluate Changes in Metabolic Markers | 30 days
  Assess the change in SCFA (namely acetate, propionate, and butyrate) production potential from baseline to 30 days.
Evaluate Changes in Inflammation Markers | 30 days
  Evaluation of the change in gut inflammatory markers (e.g., hexa-LPS Index, mucus degradation species, hydrogen sulfide levels) between at baseline and at 30 days to investigate potential anti-inflammatory effects of HMO supplementation.

CONTACTS AND LOCATIONS:
Locations (1):
- Seeding Inc, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No